CLINICAL TRIAL: NCT01908192
Title: An Adaptive, Phase IIb/III, Double-Blind, Randomized, Placebo-Controlled, Multi-Center Study of the Safety and Efficacy OF NaBen® , A D-Amino Acid Oxidase Inhibitor, as an Add-on Treatment for Schizophrenia in Adolescents
Brief Title: Adaptive Phase II Study to Evaluate the Safety & Efficacy of NaBen®
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: SyneuRx International (Taiwan) Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNR-01-NaBen
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Schizophrenia
Keywords: Sodium Benzoate; Schizophrenia; Adolescent; Antipsychotic; Anti-psychotic; NMDA; NaBen; pediatric
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NaBen® (Experimental): NaBen® is a white oral tablet (500 mg), which will be taken twice daily at a total dose of 1000 mg/day during this study.
  Interventions: Drug: NaBen®
- Placebo (Placebo Comparator): The control treatment is placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NaBen® — The Study Treatment is NaBen®, which will look, and will be packaged and maintained exactly the same way as the Control Treatment (Placebo).
  Arms: NaBen®
Drug: Placebo — The ingredients in the Control Treatment are exactly the same as in the Study Treatment, except without the primary active ingredient.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if NaBen® is a safe and effective add-on treatment for schizophrenia in adolescents.

DETAILED DESCRIPTION:
This is a two-part, multi-center, prospective, randomized, placebo-controlled, parallel-group study, in which adolescent subjects with schizophrenia will be enrolled. Overall, eligible subjects will be randomized in a pre-defined 1:1 ratio to NaBen® or placebo.

This study will be conducted in two parts:

In Part 1 (Phase IIb) of the study, 76 subjects (~ 60% of the total planned subjects) will be randomized in a 1:1 ratio (NaBen® or placebo), of which 38 subjects will be randomized to the NaBen® group and 38 subjects to the placebo group. An interim analysis (IA) will be conducted after the randomization of the 76th subject in Part 1 of the study. The data will be analyzed after all enrolled subjects in Part 1 of the study complete Visit 5 (week 6) or are withdrawn from the study, whichever occurs first. The data from IA will be reviewed by an independent Data Safety and Monitoring Committee (DSMC) that will be responsible for the review of the data from the Part 1 (Phase IIb) of the study for both safety and the effectiveness.

In Part 2 (Phase III) of the study, a total of 50 subjects will be randomized, of which 25 subjects will be randomized to the NaBen® group and 25 subjects to the placebo group. The final subject numbers in the study will depend on the sample size re-estimation after Part 1 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are between 12 and 17 years of age inclusive
* Physician confirmed DSM-IV or -V diagnosis of schizophrenia based on MINI International Neuropsychiatric Interview for Schizophrenia and Psychotic Disorders Studies for Children and Adolescents, version 6.0 (MINI-KID, Version 6.0)
* Are clinically stable with residual symptoms, defined as a total score of ≥ 60 of PANSS and a score of ≥ 40 for SANS
* An unchanged antipsychotic medication regimen for at least eight (8) weeks prior to randomization into the study and expected to remain unchanged during the study (longer for depot or long-acting antipsychotics: ten (10) months for Aripiprazole (Maintena®) and Paliperidone (Xeplion®); six (6) months for Olanzapine pamoate monohydrate (Zypadhera®); and at least 6 times duration of the reported half life or minimum four (4) months for other depot or long-acting antipsychotics)
* In good general physical health and all physical exam, neurological exam and laboratory assessments (urine/blood routine, biochemical tests and ECG) are clinically unremarkable per the investigator
* Subject has a negative urine illicit drug screening test
* Subject understands and is willing to sign the Informed Assent Form (IAF) prior to study entry and agrees to be available for all the study visits
* The subject's guardian understands and is willing to sign the Informed Consent Form (ICF) prior to study entry and agrees to be available for all the study visits
* Must not be a danger to self or others and must have family support available to be maintained as outpatients

Exclusion Criteria:

* Meets the DSM-IV or -V criteria at screening for mental retardation, dissociative disorder, bipolar disorder, major depressive disorder, schizoaffective disorder, schizophreniform disorder, autistic disorder, or primary substance induced psychotic disorder. Other comorbid disorders; e.g., attention-deficit hyperactivity disorder (ADHD), are allowed as long as schizophrenia is the primary diagnosis and the comorbid disorder(s) do not require medication.
* Subjects whose illness was resistant to antipsychotics according to prior trials of two different antipsychotics of adequate dose
* History of epilepsy, head trauma, or neurological illness other than Tourette's syndrome
* History of allergic reaction to sodium benzoate
* Serious medical illnesses such as acute or chronic renal disease, liver failure or heart disease that, in the opinion of the investigator, may interfere with the conduct of the study.
* Current substance abuse or positive urine illicit drug screening or history of substance dependence (including alcohol, but excluding nicotine and caffeine) in the past three (3) months.
* Use of depot antipsychotics in the past six (6) months
* Inability to follow protocol
* Body Mass Index (BMI) > 35
* Female subjects who are pregnant (as confirmed by urine pregnancy test performed at screening Visit) or are nursing, or who do not agree to abstinence or birth control during the study
* Cancer within the last three (3) years except for basal cell carcinoma and squamous cell carcinoma
* Previous participation in an intervention trial within 30 days of randomization
* Subjects whose PANSS score has decreased more than 10 percent during the Screening Phase

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in Positive and Negative Syndrome Scale (PANSS) total score after 6 weeks of treatment | Positive and Negative Syndrome Scale will be assessed at Visit 1 (Screening), Visit 3, 4, 5, and 6.

SECONDARY OUTCOMES:
Percent change from baseline in Positive and Negative Syndrome Scale (PANSS) total score from baseline after 6 weeks of treatment | Positive and Negative Syndrome Scale will be assessed at Visit 1 (Screening), Visit 3, 4, 5, and 6.
Percentage of subjects with 20% or more reduction in Positive and Negative Syndrome Scale (PANSS) total score from baseline after six (6) weeks of treatment | Positive and Negative Syndrome Scale will be assessed at Visit 1 (Screening), Visit 3, 4, 5, and 6
Percent change in Positive and Negative Syndrome Scale (PANSS) sub-scales | Positive and Negative Syndrome Scale will be assessed at Visit 1 (Screening), Visit 3, 4, 5, and 6.
Percent change in Scale for Assessment of Negative Symptoms (SANS) total scores | Scale for Assessment of Negative Symptoms will be assessed at Visit 1 (Screening), Visit 3,4,5, and 6
Percent change in Scale for Assessment of Negative Symptoms (SANS) sub-scale scores | Scale for Assessment of Negative Symptoms will be assessed at Visit 1 (Screening), Visit 3,4,5, and 6
Percent change from baseline in the PANSS total score after 6 weeks of treatment | Positive and Negative Syndrome Scale will be assessed at Visit 1 (Screening), Visit 3, 4, 5, and 6

OTHER OUTCOMES:
Percent change in Children's Global Assessment Scale (CGAS) | Children's Global Assessment Scale will be assessed at Visit 1(Screening), Visit 3, 4, 5, and 6
Percent change in Clinical Global Impression-Severity (CGI-S) | Clinical Global Impression will be assessed at Visit 1 (Screening), Visit 3, 4, 5, and 6
Percent change in Children's Depression Rating Scale-Revised (CDRS-R) | Children's Depression Rating Scale will be assessed at Visit 1 (Screening), Visit 3, 4, 5, and 6

CONTACTS AND LOCATIONS:
Overall Officials: Robert Findling, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (23):
- United States (20):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - CiTrials, Bellflower, California
  - Renew Behavioral Health, Inc., Long Beach, California
  - CiTrials, Riverside, California
  - Institute of Living/Hartford Hospital, Hartford, Connecticut
  - Children's National Health System, Washington D.C., District of Columbia
  - Premier Clinical Research Institute, Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - John Hopkins University - Hugo W Moser Research Institute at Kennedy Krieger Inc., Baltimore, Maryland
  - University of Massachusetts Medical School - Psychiatry Department, Worcester, Massachusetts
  - Michigan Clinical Research Institute, Ann Arbor, Michigan
  - University of Minnesota Medical Center - Department of Psychiatry, Minneapolis, Minnesota
  - Precise Research Centers, Flowood, Mississippi
  - Finger Lakes Clinical Research, Rochester, New York
  - University of Cincinnati - Dept. of Psychiatry and Behavioral Neuroscience, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Focus and Balance LLC, San Antonio, Texas
  - Pacific Institute of Medical Sciences, Bothell, Washington
  - Zain Research, LLC, Richland, Washington
- Taiwan (3):
  - Chang Gung Memorial Hospital (Linkou), New Taipei City
  - Chang Gung Memorial Hospital (Taipei), Taipei
  - Veteran General Hospital Taipei, Taipei

REFERENCES:
- See also: The clinical trial management organization — http://www.amarexcro.com
- See also: Sponsor — http://www.syneurx.com
- See also: Trial Background — http://syneurx.net